CLINICAL TRIAL: NCT04200885
Title: Comparison Of The Effectiveness Of Submucosal Corticosteroid Injection And Elastic Therapeutic Bandage Applications On Pain, Swelling And Trismus After Surgical Removal Of Mandibular Third Molar Teeth
Brief Title: Is Therapeutic Elastic Bandage As Effective As Corticosteroids Following Third Molar Surgery?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Aras Erdil, Research Assistant, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-KAEK-100
Record Dates: First submitted 2019-12-08; First posted 2019-12-16 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Third Molar Surgery
Keywords: Dexamethasone; Applied Kinesiology; Non-Steroidal Anti-Inflammatory Agents; Teeth, Impacted; Edema; Trismus; Postoperative Pain
MeSH Terms: conditions — Tooth, Impacted; Edema; Trismus; Pain, Postoperative | interventions — dexketoprofen trometamol; dexamethasone 21-phosphate; Injections, Intramuscular

STUDY DESIGN:
Intervention Model Description: Among the patients randomized because of severe postoperative sequelae expected as a result of radiological examination prior to surgical extraction of lower third molar teeth; postoperatively nonsteroid antiinflammatory drug prescribed group compared with preoperative single dose intraoral submucosal corticosteroid administration and postoperative therapeutic elastic bandage application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Postoperative NSAID Prescription (Active Comparator): Patients in this arm received common postoperative prescriptions following removal of their impacted third molars for seven days; twice a day 500 mg amoxicillin+125 mg clavulanic acid, twice a day 25 mg dexketoprofen trometamol and three times a day 1.5 mg/ml clorhexidine gluconate+1.2 mg/ml benzydamine hydrochloride containing 200 ml mouthwash.
  Interventions: Drug: Dexketoprofen Trometamol
- Preoperative Submucosal Corticosteroid Injection (Active Comparator): Patients in this arm were administered 8mg/2ml dexamethasone 21-phosphate preoperatively after local anesthesia were obtained. Injection site was the depth of buccal sulcus near operation site. For the patients in this arm 25 mg dexketoprofen trometamol was excluded from postoperative prescription in order not to affect the anti-inflammatory effects of corticosteroid. Instead of NSAID, three times a day 500 mg paracetamol was prescribed. The patients were advised not to exceed maximal dosage of 3000 mg (6 tablets) in a day.
  Interventions: Drug: Dexamethasone 21-Phosphate
- Postoperative Therapeutic Elastic Bandage Application (Active Comparator): In this arm the therapeutic elastic bandage applications were immediately performed after removal of mandibular third molars. The distance between tragus-lateral commissura line and supraclavicular lymph nodes was measured and the tapes were then cut into 5 tails. The base of the tape was placed on supraclavicular lymph nodes and tails were placed on the site to cover parotid, submandibular, submental and superficial cervical lymph nodes. The tapes were removed on postoperative second day.
  Interventions: Device: Therapeutic Elastic Bandage

INTERVENTIONS:
Drug: Dexketoprofen Trometamol — Patients were instructed to record the number of drugs they used until the second and seventh postoperative days.
  Other Names: Arveles 25 mg 20 tablets
  Arms: Postoperative NSAID Prescription
Drug: Dexamethasone 21-Phosphate — Injections were administered in the immediate preoperative period as a single shot.
  Other Names: Dekort 8mg/2ml Intramuscular (IM)/ Intravenous (IV)
  Arms: Preoperative Submucosal Corticosteroid Injection
Device: Therapeutic Elastic Bandage — The bands' lengths were individually measured and divided into five equal parts up to 2/3 of their lengths to obtain fan-type shape.
  Other Names: Kinesio Tex Gold Fingerprint (FP)
  Arms: Postoperative Therapeutic Elastic Bandage Application

SUMMARY:
In this study; Among the patients randomized because of severe postoperative sequelae expected as a result of radiological and clinical examinations; nonsteroid antiinflammatory drug prescribed group compared with preoperative single dose intraoral submucosal corticosteroid administration and therapeutic elastic bandage application considering inflammatory symptoms' severity and health related quality of life following surgical removal of impacted third molars. The study hypothesis was formed stating that corticosteroid injection and elastic bandage application would reduce the inflammatory symptoms more than NSAID.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years
* American Society of Anesthesiologists (ASA) Class 1 physiological status
* Consistent radiological and clinical data
* Volunteered to participate in the study
* Surgical difficulty score above 5 which was determined according to Pederson scale.

Exclusion Criteria:

* Being out of age range
* Analgesic or antibiotic therapy history in last 30 days due to symptoms of related third molar
* Smoking cigarette
* Any pathology associated with impacted third molar
* Active complaints on preoperative examination on the day of surgery
* Immunosuppressed or diagnosed with malignancy
* Diagnosed chronic diseases such as; Diabetes mellitus (DM), hypertension, cerebrovascular event, psychiatric diseases, coagulopathies
* Autoimmune diseases
* If total operation time exceeds 45 minutes
* Patients who could not attend regular follow-up visits
* Allergy to the medications prescribed or utilized in study protocol
* Inconsistent clinical and radiological data

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
Preoperative Pain Intensity | On the day of surgery preoperatively
  The patients were asked to mark their pain intensities on a Numerical Rating Scale in which '0' means no pain, '5' means moderate pain and '10' means worst imaginable pain on the day of surgery preoperatively.
Change From Baseline Maximal Mouth Opening on Postoperative Follow Up Visits | Preoperatively on the day of surgery, postoperative second and seventh days.
  All patients' maximal mouth opening were measured and recorded as the distance between upper and lower right central incisors.
Change From Baseline Facial Measurements on Postoperative Follow Up Visits | Preoperatively on the day of surgery, postoperative second and seventh days.
  Measurements were performed on the ipsilateral site between tragus and lateral commissura, lateral canthus and angle of mandible with a flexible ruler. The obtained values' average amounts were calculated and recorded for each patient.
Oral Analgesic Consumption-1 | Postoperative Second Day
  The patients were asked to record the amounts of consumed analgesic tablets (tablets per day) until first follow up visit.
Postoperative Pain Intensity-1 | Postoperative Second Day
  The patients were asked to mark their pain intensities on a Numerical Rating Scale in which '0' means no pain, '5' means moderate pain and '10' means worst imaginable pain.
Postoperative Pain Intensity-2 | Postoperative Seventh Day
  The patients were asked to mark their pain intensities on a Numerical Rating Scale in which '0' means no pain, '5' means moderate pain and '10' means worst imaginable pain.
Oral Analgesic Consumption-2 | Postoperative Seventh Day
  The patients were asked to record the amounts of consumed analgesic tablets (tablets per day) between first and last follow up visits.

SECONDARY OUTCOMES:
Wound Healing Scores | Postoperative second and seventh days.
  Extraction wound healing rates were evaluated by Landry's healing index. The index scores were classified as; 1. Very poor, 2. Poor, 3. Good, 4. Very Good and 5. Excellent.
Oral Health Impact Profile | Preoperatively on the day of surgery, postoperative second and seventh days.
  Oral health-related quality of life was followed up with Oral Health Impaction Profile-14 questionnaire (Turkish Version). The investigators aimed to detect the alterations in quality of life due to surgical intervention and the other treatment modalities. The obtainable scores vary between 0-56 points. Lower scores indicate better postoperative physical and psychological conditions.
Postoperative Symptom Severity Evaluation | Postoperative seventh day.
  Postoperative inflammatory symptoms were evaluated with the postoperative symptom severity scale at the end of the follow-up period individually. The scale scores vary between 0%-100%. The higher scores indicate that the individual experienced severe symptoms. The investigators aimed to detect the severity of symptoms from the point of the patient's view.

CONTACTS AND LOCATIONS:
Overall Officials: Nihat Akbulut, Assoc. Dr., Study Director — Tokat Gaziosmanpasa University
Locations (1):
- Tokat Gaziosmanpasa University, Faculty of Dentistry, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) related to study protocol and results will be shared during submitting as an article.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The study will be transformed to an article in six months.
Access Criteria: All IPD and supporting information data will be accessible after publication of the article

REFERENCES:
- [Background] Ristow O, Hohlweg-Majert B, Sturzenbaum SR, Kehl V, Koerdt S, Hahnefeld L, Pautke C. Therapeutic elastic tape reduces morbidity after wisdom teeth removal--a clinical trial. Clin Oral Investig. 2014 May;18(4):1205-1212. doi: 10.1007/s00784-013-1067-3. Epub 2013 Aug 21. PMID 23963616
- [Background] Alcantara CE, Falci SG, Oliveira-Ferreira F, Santos CR, Pinheiro ML. Pre-emptive effect of dexamethasone and methylprednisolone on pain, swelling, and trismus after third molar surgery: a split-mouth randomized triple-blind clinical trial. Int J Oral Maxillofac Surg. 2014 Jan;43(1):93-8. doi: 10.1016/j.ijom.2013.05.016. Epub 2013 Jun 28. PMID 23810681
- [Background] Deo SP. Single-Dose of Submucosal Injection of Dexamethasone Affects the Post Operative Quality of Life After Third Molar Surgery. J Maxillofac Oral Surg. 2016 Sep;15(3):367-375. doi: 10.1007/s12663-015-0846-6. Epub 2015 Dec 7. PMID 27752209
- [Derived] Erdil A, Akbulut N, Altan A, Demirsoy MS. Comparison of the effect of therapeutic elastic bandage, submucosal dexamethasone, or dexketoprofen trometamol on inflammatory symptoms and quality of life following third molar surgery: a randomized clinical trial. Clin Oral Investig. 2021 Apr;25(4):1849-1857. doi: 10.1007/s00784-020-03487-y. Epub 2020 Aug 15. PMID 32803439